CLINICAL TRIAL: NCT03858556
Title: Prospective Observation Study of the Effect of Chuna Manipulation Therapy on Gait in Patients With Lumbar Disc Herniation
Brief Title: Effect of Chuna Manipulation Therapy on Gait in Patients With Lumbar Disc Herniation
Status: Withdrawn | Type: Observational
Why Stopped: Study plan was changed, this project would not be in progress
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2018-08 Gait analysis
Record Dates: First submitted 2018-12-17; First posted 2019-02-28 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-02

CONDITIONS: Lumbar Disc Herniation; Gait Analysis; Manual Therapy
Keywords: gait; effectiveness; treatment; Lumbar intervertebral disc herniation; Chuna
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Phytotherapy; Acupuncture Therapy; Electroacupuncture; Cupping Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with lumbar disc herniation: 3times(baseline, 1weeks, 2weeks) of Observation of gait, Oswestry disability index, EQ5D-5L, Lumbar Range of motion in inpatients with lumbar intervertebral disc herniation hospitalized at Korean medicine hospital.
  -Integrative Korean medicine treatment Procedure/Surgery: Chuna manipulation Drug: Herbal medicine Procedure/Surgery: Bee venom pharmacopuncture Procedure/Surgery: Pharmacopuncture Procedure/Surgery: Acupuncture Procedure/Surgery: Electroacupuncture Procedure/Surgery: Cupping Other intervention(s) Other: Other intervention(s)
  Interventions: Procedure: Chuna manipulation; Drug: Herbal medicine; Procedure: Bee venom pharmacopuncture; Procedure: Pharmacopuncture; Procedure: Acupuncture; Procedure: Electroacupuncture; Procedure: Cupping; Other: Other intervention(s)
- Normal: baseline Observation of gait, Oswestry disability index, EQ5D-5L, Lumbar Range of motion.
  -No treatment

INTERVENTIONS:
Procedure: Chuna manipulation — Chuna is a Korean spinal manipulation that incorporates spinal manipulation techniques for joint mobilization involving high-velocity, low amplitude thrusts to joints slightly beyond the passive range of motion and gentle force to joints within the passive range of movement. Chuna manipulation will be administered to pelvic, lumbar, thoracic, and cervical vertebrae at the physician's discretion.
  Other Names: Chuna spinal manipulation
  Groups: Patients with lumbar disc herniation
Drug: Herbal medicine — Herbal medicine will be administered in water-based decoction (120ml) and dried powder (2g) form (Ostericum koreanum, Eucommia ulmoides, Acanthopanax sessiliflorus, Achyranthes japonica, Psoralea corylifolia, Saposhnikovia divaricata, Cibotium barometz, Lycium chinense, Boschniakia rossica, Cuscuta chinensis, Glycine max, Atractylodes japonica).
  Other Names: Traditional herbal medicine
  Groups: Patients with lumbar disc herniation
Procedure: Bee venom pharmacopuncture — Bee venom pharmacopuncture will be administered only after confirming a negative response to hypersensitivity skin test. Diluted bee venom (saline:bee venom ratio, 10,000:1) filtered for allergens will be injected at 4-5 acupoints proximal to the dysfunctional site at the physician's discretion. Each acupuncture point will be injected to a total of 0.5-1 cc using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea).
  Other Names: Bee venom acupuncture
  Groups: Patients with lumbar disc herniation
Procedure: Pharmacopuncture — Pharmacopuncture consisting of select herbal ingredients will be administered at Hyeopcheok (Huatuo Jiaji, EX B2), Ah-shi points and local acupuncture points using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea).
  Groups: Patients with lumbar disc herniation
Procedure: Acupuncture — Acupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
  Groups: Patients with lumbar disc herniation
Procedure: Electroacupuncture — Electroacupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
  Groups: Patients with lumbar disc herniation
Procedure: Cupping — Cupping treatment will be administered at 1-2 points using mainly proximal acupuncture points and Ah-shi points.
  Groups: Patients with lumbar disc herniation
Other: Other intervention(s) — Patients will be allowed any other additional intervention(s) as deemed necessary by the attending physician regardless of type or dose, and patterns of use will be investigated and recorded as an pragmatic clinical study.
  Groups: Patients with lumbar disc herniation

SUMMARY:
Prospective Observation Study of the Effect of Chuna Manipulation Therapy on Gait in Patients With Lumbar Disc Herniation

DETAILED DESCRIPTION:
To investigate the effect of Chuna manual therapy on gate, 20 patients with lumbar disc herniation were studied. The gait analysis was performed before the first treatment, after the seventh treatment, after the 14th treatment, and compared with the data of 20 normal subjects.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar intervertebral disc herniation as confirmed by a doctor of medicine or a doctor of Korean medicine through an MRI
* Patients with radiculopathy
* Patients aged 19 to 60
* Patients with an Oswestry Disability Index (ODI) of ≥10
* Patients who have agreed to participate in the clinical study and given written informed consent

Exclusion Criteria:

* Patients who were unable to walk for more than 5 minutes due to pain
* Patients with a serious disease that may limit gait(such as spinal metastasis of the tumor, acute fracture and spinal dislocation)
* Patients with chronic conditions that may interfere with the interpretation of the therapeutic effect or outcome(such as chronic kidney failure)
* Patients with progressive neurological deficit or severe neurological symptoms such as spinal cord injury
* Patients with severe mental illness
* Patients who are currently on on steroids, immunosuppressants, psychiatric medications, or other medications that can affect outcome
* Patients who are pregnant or planning a pregnancy
* Patients who are participating in other clinical studies or if it is difficult for you to participate in clinical research as determined by the researcher

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who are admitted to Jaseng Hospital of Korean Medicine
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Gait parameter change | baseline, 2 weeks after baseline
  - Time parameters(step time)

SECONDARY OUTCOMES:
ODI | baseline, 2 weeks after baseline
  Oswestry Disability Index(ODI)
EQ-5D | baseline, 2 weeks after baseline
  EuroQol-5 Dimension(EQ-5D)
Lumbar ROM | baseline, 2 weeks after baseline
  Lumbar Range of Motion(ROM) (Flexion/Extension/Lateral flexion/Rotation)
SLR | baseline, 2 weeks after baseline
  Straight Leg Raise test(SLR)

IPD SHARING:
Plan to Share IPD: No